CLINICAL TRIAL: NCT06116864
Title: Enhancing Polyp Detection: A Randomized Controlled Trial Comparing Combined Computer-Aid Detection and Polyp-Detecting Colonoscope Attachment to Computer-Aid Detection Alone in Patients Undergoing Colonoscopy.
Brief Title: Enchasing Polyp Detection: The Effect of Adding Polyp Detection Attachment Device to Computer Aid Detection System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Wesam Frandah, Associate Professor, Marshall University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2094805
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Colon Cancer Screening; Colon Cancer Surveillance
Keywords: Colon cancer screening; Colon cancer surveillance; Computer-Aided Detection of adenoma; Colonoscope attachment device; Endocuff

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial that compares Endocuff with Gi Genius (group A) to GI Genius alone (group B) for patients who are undergoing elective outpatient colonoscopy. Patients will be randomized by a secure online randomization software that will allocate patients in a 1:1 ratio to group A or group B.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Endocuff + GI Genius (Experimental): Endocuff is a polyp-detecting colonoscope attachment device. GI Genius is and Computer-Aid Detection (CADe) system to detect polyps
  Interventions: Device: Endocuff and GI Genius
- GI Genius (Active Comparator): GI Genius is and Computer-Aid Detection (CADe) system to detect polyps
  Interventions: Device: GI Genius

INTERVENTIONS:
Device: Endocuff and GI Genius — Endocuff is a polyp-detecting colonoscope attachment device. GI Genius is and Computer-Aid Detection (CADe) system to detect polyps
  Arms: Endocuff + GI Genius
Device: GI Genius — GI Genius is and Computer-Aid Detection (CADe) system to detect polyps
  Arms: GI Genius

SUMMARY:
Despite the widespread use of colonoscopy, the ongoing challenge of potentially missing polyps remains. Previous studies have independently shown that both Endocuff, a colonoscope attachment device for polyp detection, and Computer-Aided Detection (CADe) systems have individually demonstrated enhanced lesion detection and safety. This study seeks to evaluate the efficacy of combining the Endocuff CADe versus using CADe alone in colonoscopy procedures for colorectal cancer screening and surveillance. This research project aims to ascertain whether the synergistic application of these technologies yields superior outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients scheduled for an outpatient screening or surveillance colonoscopy.

Exclusion Criteria:

* Patients who require diagnostic colonoscopy (e.g.; anemia or GI bleeding).
* Patients requiring deep ileal intubation.
* Patients with inflammatory bowel disease.
* Patients with radiotherapy-induced colitis or other severe colitis.
* Patients with colonic strictures.
* Patients with acute diverticulitis.
* Patients with large bowel obstruction.
* Patients scheduled for therapeutic colonoscopy (e.g., planned endoscopic mucosal resection for known polyps).
* Patients scheduled for assessment of a known colonic lesion.
* Patients with a known history of hereditary polyposis syndrome or untreated colon cancer.
* Patients with a history of colon resection.
* Patients on continuous anti-thrombotic therapy
* Pregnancy.
* Patients who are ineligible for colonoscopy due to medical or psychiatric conditions.
* Patients who are vulnerable or unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1766 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 18 months
  It is the percentage of patients who have at least one adenoma detected during the colonoscopy

SECONDARY OUTCOMES:
Polyp detection rate | 18 months
Number of cancerous lesions | 18 months
Differences in polyps histology between the groups | 18 months
Differences in polyps size | 18 months
Polyps location (cecum, ascending, transverse, descending, sigmoid, or rectum) | 18 months
Cecal intubation rate | 18 months
Cecal intubation time | 18 months
Colonoscopy withdrawal time | 18 months
Procedure complication (bleeding or perforation) by the end of the procedure. (Following lexicon for endoscopic adverse events methods) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Wesam Frandah, MD, Principal Investigator — Marshall University Joan C. Edwards School of Medicine
Locations (1):
- Marshall University Joan C. Edwards School of Medicine/Cabell Huntington Hospital, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No